CLINICAL TRIAL: NCT02768753
Title: Comparison Between the Axillary Bilateral-breast Approach (ABBA) and Bilateral Axillo-breast Approach (BABA) for Robotic Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jinan Military General Hospital (Other)
Responsible Party: Principal Investigator, Gaofeng Ni, Resident Doctor, Jinan Military General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ShandongJJZY-01
Record Dates: First submitted 2016-05-02; First posted 2016-05-11 (Estimated); Results first posted 2019-09-27 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Thyroid Papillary Carcinoma; Thyroidectomy
Keywords: Robotic thyroidectomy; Robotic central neck dissection; Axillary bilateral-breast approach; Bilateral axillo-breast approach
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- The Axillary Bilateral-breast Approach (ABBA) group (Experimental): All patients were told about the operative techniques involved in robotic thyroidectomy via the Axillary Bilateral-breast Approach (ABBA) and Bilateral Axillo-breast Approach (BABA), and patients subsequently chose their preferred surgical procedure, voluntarily agreed to participate in our study, and provided written informed consent.
  Interventions: Procedure: The Axillary Bilateral-breast Approach
- The bilateral Axillo-breast Approach (BABA) group (Experimental): All patients were told about the operative techniques involved in robotic thyroidectomy via the Axillary Bilateral-breast Approach (ABBA) and Bilateral Axillo-breast Approach (BABA), and patients subsequently chose their preferred surgical procedure, voluntarily agreed to participate in our study, and provided written informed consent.
  Interventions: Procedure: The bilateral Axillo-breast Approach

INTERVENTIONS:
Procedure: The Axillary Bilateral-breast Approach
  Arms: The Axillary Bilateral-breast Approach (ABBA) group
Procedure: The bilateral Axillo-breast Approach
  Arms: The bilateral Axillo-breast Approach (BABA) group

SUMMARY:
The purpose of this study is to compare the therapeutic effects between the axillary bilateral-breast approach (ABBA) and bilateral axillo-breast approach (BABA) for robotic thyroidectomy.To explore the efficacy, safety, cosmetic results and clinical value by the two approaches.

DETAILED DESCRIPTION:
Although several reports on operative outcomes of the robotic technique have appeared, no prospective trials comparing the clinical results of between the axillary bilateral-breast approach (ABBA) and bilateral axillo-breast approach (BABA) for robotic thyroidectomy have been described. The investigators therefore designed a prospective trial comparing outcomes, including surgical outcomes and patient satisfaction, between patients undergoing robotic and conventional open thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

1. the initial surgery
2. preoperative needle aspiration biopsy of thyroid cancer, and the diameter of no more than 1cm, no lateral neck lymph node metastasis
3. the tumor is confined to the thyroid membrane, not invading trachea and recurrent laryngeal nerve
4. intraoperative frozen section diagnosis of thyroid cancer
5. the patient informed consent.

Exclusion Criteria:

1. high-frequency ultrasound preoperative tumor diameter greater than 1cm, or lateral neck lymph node metastasis in patients
2. there had been a history of thyroid surgery or neck radiation therapy
3. pregnant or lactating women
4. with severe Hashimoto's thyroiditis, thyroid volume greater than II °
5. coagulation disorders, hyperthyroidism or hypothyroidism patients
6. sternal goiter.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of thyroid and breast surgery, General Hospital of Jinan Military Area, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- The Axillary Bilateral-breast Approach (ABBA) Group: All patients were told about the operative techniques involved in robotic thyroidectomy via the Axillary Bilateral-breast Approach (ABBA) and Bilateral Axillo-breast Approach (BABA), and patients subsequently chose their preferred surgical procedure, voluntarily agreed to participate in our study, and provided written informed consent.
  The Axillary Bilateral-breast Approach
- The Bilateral Axillo-breast Approach (BABA) Group: All patients were told about the operative techniques involved in robotic thyroidectomy via the Axillary Bilateral-breast Approach (ABBA) and Bilateral Axillo-breast Approach (BABA), and patients subsequently chose their preferred surgical procedure, voluntarily agreed to participate in our study, and provided written informed consent.
  The bilateral Axillo-breast Approach
Period: Overall Study
Arm/Group | The Axillary Bilateral-breast Approach (ABBA) Group | The Bilateral Axillo-breast Approach (BABA) Group
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | The Axillary Bilateral-breast Approach (ABBA) Group | The Bilateral Axillo-breast Approach (BABA) Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.30 (10.95) | 38.20 (9.82) | 41.25 (10.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 22 | 25 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 30 | 30 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index（BMI） [Mean (Standard Deviation); unit: kg / m ^ 2] — units:kg / m ^ 2 Mean(Standard Deviation)
  kg / m ^ 2 | 22.92 (3.54) | 23.64 (3.21) | 23.28 (3.37)

OUTCOME MEASURES:

1. Primary Outcome: Change of VAS Pain Scores for the First 24 Hours
Description: The visual analogue scale is utilized to assess the postoperative pain change for the first 24 hours.Using a 10cm straight line, one end is marked 0 for "pain free" and the other end is marked 10 for "unbearable pain". The pain intensity of the patient's own feelings was marked on a straight line, and the length from 0 to the marked point represented the pain level of the patient. The evaluation criteria of VAS were as follows: 0 for pain, 3 for mild pain, 4 to 6 for moderate pain and 7 to 10 for severe pain.Lower values represent better outcomes, higher values represent worse outcomes.
Time Frame: The pain scores of 2pm, 10pm and 6am on the first day after operation were evaluated.The mean values were calculated and recorded.
Measure: Mean (Standard Deviation); unit: score
Arm/Group | The Axillary Bilateral-breast Approach (ABBA) Group | The Bilateral Axillo-breast Approach (BABA) Group
Number analyzed (Participants) | 30 | 30
score | 2.13 (1.10) | 2.33 (1.34)

2. Primary Outcome: Cosmetic Outcomes
Description: The satisfaction with cosmetic outcomes was analyzed quantitatively using a scoring system that ranged from 1 to 4(1, extremely; 2, fairly; 3, normal; 4: not at all) that was rated by patients at the outpatient clinic 3 months after the operation.
Time Frame: 3 months after surgery
Measure: Mean (Standard Deviation); unit: score
Arm/Group | The Axillary Bilateral-breast Approach (ABBA) Group | The Bilateral Axillo-breast Approach (BABA) Group
Number analyzed (Participants) | 30 | 30
score | 3.17 (0.93) | 3.90 (0.31)

3. Secondary Outcome: Subjective Voice
Description: We have developed a questionnaire with a total of 30 questions, each with a score of 4, and the patients scored according to their own situation. The highest score of the questionnaire is 120, the lowest score is 0, the best, the score is 0-30, 30-60 is good, 60-90 is normal, 90-120 is poor.
Time Frame: After operation 8 a.m. on the 7th day
Measure: Mean (Standard Deviation); unit: score
Arm/Group | The Axillary Bilateral-breast Approach (ABBA) Group | The Bilateral Axillo-breast Approach (BABA) Group
Number analyzed (Participants) | 30 | 30
score | 10.27 (3.77) | 10.70 (2.69)

4. Secondary Outcome: Swallowing Evaluation
Description: The patient sat upright and drank 30 ml warm boiled water to observe the time required and the cough.
  1. score (excellent) can swallow water smoothly once
  2. score (good) more than 2 times, can swallow without coughing
  3. score (middle) can swallow once, but have a choking cough
  4. score (may) more than 2 times swallowing, but with choking cough
  5. score (difference) frequent cough, not all swallowing Calculate the average value for statistical analysis
Time Frame: 8 a.m. on the 3rd day after operation
Measure: Mean (Standard Deviation); unit: score
Arm/Group | The Axillary Bilateral-breast Approach (ABBA) Group | The Bilateral Axillo-breast Approach (BABA) Group
Number analyzed (Participants) | 30 | 30
score | 1.23 (0.43) | 1.27 (0.45)

ADVERSE EVENTS:
Time Frame: From the beginning of the operation to 1 years after the operation
Description: First of all, our operation team has a very rich experience in thyroid surgery(More than 120 cases of thyroid surgery by Da VinciSi have been successfully implemented). Secondly, we are using the Da VinciSi strictly.
Arm/Group | The Axillary Bilateral-breast Approach (ABBA) Group | The Bilateral Axillo-breast Approach (BABA) Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-04-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT02768753/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT02768753/SAP_001.pdf